CLINICAL TRIAL: NCT04872556
Title: Evaluation of the Effect of Laser Acupuncture on Myalgia and Arthralgia During Docetaxel or Paclitaxel Treatment in Cancer Patients
Brief Title: Evaluation of the Effect of Laser Acupuncture on Taxane Acute Pain Syndrome Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: end of the supporting fund
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202001710A3
Record Dates: First submitted 2021-04-21; First posted 2021-05-04 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2021-03

CONDITIONS: Pain Cancer; Joint Pain
Keywords: Laser acupuncture; Taxanes; Chemotherapy; Cancer; Myalgia; Arthralgia
MeSH Terms: conditions — Cancer Pain; Arthralgia; Neoplasms; Myalgia

STUDY DESIGN:
Intervention Model Description: Participants would be 90 cancer patients accepted Taxanes treatment who are suffered from myalgia and Arthralgia. The investigators would put 45 participants in experimental groups and the other 45 participants in control group with randomization.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The investigators would put eye masking over participants. The care providers would not know the laser acupuncture device or pseudo-laser acupuncture device with randomization. The investigator did not know which group the participants belonged with.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser acupuncture group (Experimental): The experiment group would arrange laser acupuncture on day1 and day3 after Taxanes treatment, besides the control group arrange pseudo-laser acupuncture. In the mean while, blood tests were performed with the C-Reactive protein, erythrocyte sedimentation rate, Interleukin-6 for each participants. Evaluation would be records on day1, day3, and day 8 after Taxanes treatment.
  Interventions: Device: Laser acupuncture device
- Pseudo-laser acupuncture group (Sham Comparator): The experiment group would arrange laser acupuncture on day1 and day 3 after Taxanes treatment, besides the control group arrange pseudo-laser acupuncture. In the mean while, blood tests were performed with the C-Reactive protein, erythrocyte sedimentation rate, Interleukin-6 for each participants. Evaluation would be records on day1, day3, and day 8 after Taxanes treatment.
  Interventions: Device: Pseudo-laser acupuncture

INTERVENTIONS:
Device: Laser acupuncture device — The experiment group would arrange laser acupuncture on day1 and day3 after Taxanes treatment. In the mean while, blood tests were performed with the C-Reactive protein, erythrocyte sedimentation rate, Interleukin-6 for each participants. Evaluation would be records on day1, day3, and day 8 after Taxanes treatment.
  Arms: Laser acupuncture group
Device: Pseudo-laser acupuncture — The experiment group would arrange Pseudo-laser acupuncture on day1 and day3 after Taxanes treatment. In the mean while, blood tests were performed with the C-Reactive protein, erythrocyte sedimentation rate, Interleukin-6 for each participants. Evaluation would be records on day1, day3, and day 8 after Taxanes treatment.
  Arms: Pseudo-laser acupuncture group

SUMMARY:
This is a prospectively randomized and double-blinded clinical study. Cancer patients were suffered from the taxanes-induced joint pain, and would be advised to receive laser acupuncture in specific points to relieve pain. Clinical effects of analgesic changes would be evaluated before and after the intervention. The inflammation associated indices would be further analyzed to reveal the therapeutic mechanism of laser acupuncture. The laser acupuncture was expected to relief taxanes-induced adverse effects in patients and also can improve patients' life quality.

DETAILED DESCRIPTION:
The current clinical study is prospectively randomized and double-blinded, and practice in Chang Gung Memorial Hospital in Linkou, TaoYuan and Taipei branches. All 90 participants suffered from taxanes-induced myalgia and Arthralgia, and will be randomly assigned into the experimental groups (45 participants) and the control group (45 participants). The experiment group would arrange laser acupuncture on day1 and day3 after Taxanes treatment, besides the control group arrange pseudo-laser acupuncture. In the mean while, blood tests were performed with the C-Reactive protein, erythrocyte sedimentation rate, Interleukin-6 for each participants. Evaluation would be records on day1, day3, and day 8 after Taxanes treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients received taxanes treatment and complained with myalgia and Arthralgia in the first taxanes treatment course.
2. Age between 20-70 years old
3. The NRS (numerical rating scale) score of pain increased more than 2 after the treatment.
4. Both 1st and 2nd taxanes treatment with the same dose

Exclusion Criteria:

1. Receiving acupuncture or herbal medicine over past three months
2. Myalgia and arthralgia were not due to taxanes treatment such osteoarthritis or rheumatic arthritis
3. Wounds or skin infections over laser acupuncture points
4. Refuse assign information consent or follow study protocol

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
NRS on Day 1 | Day 1 after Taxanes treatment
  Numerical rating scale in pain evaluation
NRS on Day 3 | Day 3 after Taxanes treatment
  Numerical rating scale in pain evaluation
NRS on Day 8 | Day 8 after Taxanes treatment
  Numerical rating scale in pain evaluation

SECONDARY OUTCOMES:
Inflammation assessment | Day 1 and day 3
  Inflammation associated indices: C-Reactive protein
Inflammation assessment | Day 1 and day 3
  Inflammation associated indices: erythrocyte sedimentation rate
Inflammation assessment | Day 1 and day 3
  Inflammation associated indices: Interleukin-6
Functional Assessment of Cancer Therapy-General Scale on Day 1 | Day 1
  A Taxanes treatment questionnaire
Functional Assessment of Cancer Therapy-General Scale on Day 3 | Day 3
  A Taxanes treatment questionnaire
Functional Assessment of Cancer Therapy-General Scale on Day 8 | Day 8
  A Taxanes treatment questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- ChangGung Memorial Hospital, Taoyuan District, Taiwan